CLINICAL TRIAL: NCT04312984
Title: The Long Term Outcomes of Micronutrient Antioxidant Supplementation in Patients With Chronic Pancreatitis
Status: Completed | Type: Observational
Sponsor: Manchester University NHS Foundation Trust (Other Government)
Responsible Party: Sponsor
Other Study IDs: CMFT-IRAS-145239-1.8
Record Dates: First submitted 2015-04-03; First posted 2020-03-18 (Actual); Last update posted 2020-03-18 (Actual); Status verified 2020-03

CONDITIONS: Chronic Pancreatitis
MeSH Terms: conditions — Pancreatitis, Chronic

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
This is a anonymised case note study looking at the long term outcomes of patients with Chronic Pancreatitis on micro nutrient antioxidant treatment.

DETAILED DESCRIPTION:
Chronic pancreatitis is the medical term for chronic inflammation of the pancreas. This illness is associated with long-term abdominal pain. In the 1980s it was proposed that chronic pancreatitis was due to a deficiency of protective "antioxidants" in the pancreas and on this basis antioxidant therapy was introduced. This therapy was highly controversial until a large randomised trial of antioxidant therapy in chronic pancreatitis, undertaken in Manchester showed that 6 months intervention with antioxidant therapy was not associated with any change in pain score or improvement in quality of life. Antioxidant therapy is no longer used in modern day pancreatic practice.

However, as with any study, the randomised trial raised some specific questions.

First, does treatment for more than 6 months provide benefit? Second, are there disease sub-types of chronic pancreatitis where antioxidant therapy may benefit?

Given the lack of contemporary use of antioxidant therapy, this question cannot be answered in a prospective study. However, the case records of the Manchester Royal Infirmary contain information on antioxidant treatment in patients who received this therapy over a prolonged period.

Thus the aim of the present study is to review the case notes of patients given a discharge code from the Manchester Royal Infirmary of chronic pancreatitis during the period 1st January 1990 to 1st January 1998 in order to assess whether there is a record of improvement in outcome. Only the case notes will be reviewed and patients will be given an opportunity to opt out.

The study accepts the limitations of assessing pain from clinical notes but also notes that more objective findings such as development of diabetes mellitus (a long term complication of chronic pancreatitis) can be assessed from the notes.

ELIGIBILITY:
Inclusion Criteria:

* Patients with Chronic Pancreatitis treated with Long term anti-oxidants

Exclusion Criteria:

* Cancer, On trials

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed with Chronic Pancreatitis using the Zurich workshop criteria
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2015-11-30 (Actual); Primary Completion 2015-12-23 (Actual); Study Completion 2015-12-23 (Actual)

PRIMARY OUTCOMES:
Pain Relief | 10 years
Insulin Dependence | 10 years

CONTACTS AND LOCATIONS:
Overall Officials: Ajith K Siriwardena, MD FRCS, Principal Investigator — CMFT
Locations (1):
- Manchester Royal Infirmary, Manchester, United Kingdom